CLINICAL TRIAL: NCT05013242
Title: Goserline Acetate Versus Dienogest in Treatment of Pain Associated With Endometriosis
Brief Title: Goserline Acetate VS Dienogest in Endometriosi
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.19.09.791.R1
Record Dates: First submitted 2021-04-20; First posted 2021-08-19 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Goserelin; Gonadotropin-Releasing Hormone; dienogest

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group use GnRH (Active Comparator): GnRH (zoladex 3.75mg) injection once every 4 weeks
  Interventions: Drug: Zoladex
- Group use Visanne (dienogest 2mg) oral once daily for 12 weeks (Active Comparator): Visanne (dienogest 2mg) oral once daily for 12 weeks
  Interventions: Drug: Visanne

INTERVENTIONS:
Drug: Zoladex — evaluate efficacy of Zoladex in complete 12 week treatment of pain in women suffer from chronic pelvic pain diagnosed as endometriosis
  Other Names: Gnrh
  Arms: group use GnRH
Drug: Visanne — valuate efficacy of Dienogest in complete 12 week treatment of pain in women suffer from chronic pelvic pain diagnosed as endometriosis
  Other Names: Dienogest
  Arms: Group use Visanne (dienogest 2mg) oral once daily for 12 weeks

SUMMARY:
clinical trial aims to evaluate efficacy of dienogest (DNG) in comparison to goserline acetate in complete 12 week treatment of pain in women suffer from chronic pelvic pain diagnosed as endometriosis by laparoscopy and histopathology.

DETAILED DESCRIPTION:
The study will be a clinical trial study of 12-week trial of GnRH (zoladex 3.75mg) injection once every 4 weeks and Visanne (dienogest 2mg) oral once daily for 12 weeks in patients confirmed endometriosis by laparoscopic surgery.

Pretreatment assessment, the patients will be questioned about their pelvic symptoms (dysmenorrhea, nonmenstrual pelvic pain, and deep dyspareunia) after taking full history and examination , The study will investigate and evaluate possible early, long side effects and efficacy of treatment to controlling the pain.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant women confirmed to have endometriosis by histopathology and not received any hormonal treatment yet. Also, medical treatment was the proper choice for treatment of each case.

Exclusion Criteria:

* Women suspect pregnancy.
* Breast feeding women.
* Previous use of hormonal agents (progestin less than 6 months, danazol less than 3 month, oral contraceptive pills less than 1 month before screening).
* Women with other gynecological pathology interfere with treatment we will use.
* Using of corticosteroids.
* Family history of osteoporosis.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-11-25 (Estimated); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
number of patients with pain symptoms reduction | 12 week
  number of patients with endometriosis-associated pain symptoms reduction

SECONDARY OUTCOMES:
assessment change in pain severity | 12 weeks
  pain severity assessment after treatment by visual analogue scale as determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark providing a range of scores from 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Mosbah, Principal Investigator — Mansoura university faculity of medicine , obstetric and gyneclogy department
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No